CLINICAL TRIAL: NCT01659996
Title: An Immunogenicity and Safety Evaluation of Menactra® (Meningococcal [Groups A, C, Y and W-135] Polysaccharide Diphtheria Toxoid Conjugate Vaccine) When Administered to Healthy Subjects at 9 Months and Concomitantly With Pentacel® at 15 to 18 Months of Age.
Brief Title: Study of Menactra® in Healthy Subjects at 9 Months and Concomitantly With Pentacel® at 15 to 18 Months of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA55; U1111-1120-1368 (Other: WHO)
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Meningitis; Meningococcal Infection; Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae Serotype b (Hib)
Keywords: Meningitis; Meningococcal Infection; Diphtheria; Pertussis; Menactra®; Pentacel®
MeSH Terms: conditions — Meningitis; Meningococcal Infections; Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections | interventions — Meningococcal Vaccines; Tetanus Toxoid; pentacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Menactra Vaccine Group (Experimental): Participants will receive Meningococcal polysaccharide diphtheria toxoid conjugate (Menactra®) at 9 months of age and Menactra® at 15 to 18 months of age.
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate
- Menactra and Pentacel Vaccine Group (Experimental): Participants will receive Meningococcal polysaccharide diphtheria toxoid conjugate (Menactra®) at 9 months of age and Menactra® + Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed (Pentacel®) concomitantly at 15 to 18 months of age.
  Interventions: Biological: Meningococcal polysaccharide diphtheria toxoid conjugate + Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed
- Pentacel Vaccine Group (Active Comparator): Participants will receive only Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Pentacel®) at 15 to 18 months of age.
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate

INTERVENTIONS:
Biological: Meningococcal polysaccharide diphtheria toxoid conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra Vaccine Group
Biological: Meningococcal polysaccharide diphtheria toxoid conjugate + Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed — 0.5 mL, Intramuscular
  Other Names: Menactra®; Pentacel®
  Arms: Menactra and Pentacel Vaccine Group
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate — 0.5 mL, Intramuscular
  Other Names: Pentacel®
  Arms: Pentacel Vaccine Group

SUMMARY:
The aim of the study is to further characterize the safety and immunogenicity of Menactra® in the population <2 years of age when administered alone and when the second dose is administered concomitantly with the 4th dose of Pentacel®, a licensed pediatric vaccine.

Primary Objectives:

* To evaluate and compare the antibody responses to meningococcal serogroups A, C, Y, and W-135 induced by 2 injections of Menactra® in subjects aged 9 months at the first vaccination visit and 15 to 18 months at the second vaccination visit.
* To evaluate and compare the antibody responses to Pertussis (pertussis toxoid [PT], filamentous haemagglutinin [FHA] and pertactin [PRN]) antigens induced by a dose of Pentacel® when administered concomitantly with Menactra® to those elicited by a dose of Pentacel® administered alone.
* To evaluate and compare the antibody responses to polyribosylribitol phosphate (PRP), tetanus and diphtheria antigens induced by a dose of Pentacel® when administered concomitantly with Menactra® to those elicited by a dose of Pentacel® alone.

Observational Objectives:

* To describe the safety profile (immediate unsolicited AEs within 30 minutes of each trial vaccination, solicited reactions within 7 days of each vaccination, unsolicited AEs within 30 days of each vaccination, and serious adverse events [SAEs] throughout the course of the trial from Day 0 up to Day 30 after the last trial vaccination[s]) in all trial groups
* To describe the antibody responses to meningococcal serogroups A, C, Y, and W-135, measured by SBA HC, 30 days after the second Menactra® administration
* To describe the antibody responses to Pentacel® (PT, FHA, PRN, FIM, diphtheria, tetanus, polio, PRP) measured by enzyme-linked immunosorbent assay (ELISA), radioimmunoassay (RIA), or functional assays.

DETAILED DESCRIPTION:
Participants will be vaccinated according to their randomized groups at age 9 months and at age 15 to 18 months. They will undergo immunogenicity assessment and safety monitoring post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 months (249 to 305 days) for Groups 1 and 2, or 15 to 18 months (420 to 570 days) for Group 3 on the day of the first trial visit
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative
* Received 3 doses of any DTaP-containing vaccines
* Received 3 doses of a Hib-containing vaccine, or 2 doses if the subject received PRP-OMP (PedvaxHIB® or Comvax®[HepB-Hib])
* Received at least 3 doses of a CRM197-based pneumococcal conjugate vaccine (Pneumococcal conjugate vaccine [PCV] or 13-Valent pneumococcal conjugate vaccine [PCV13])
* Subject and parent/ legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding each trial vaccination or planned receipt of any vaccine in the 4 weeks following each trial vaccination, except for influenza vaccination, which may be received at least 2 weeks before or after the trial vaccination(s)
* Vaccination against meningococcal disease with either the trial vaccine or another vaccine, or receipt of the 4th dose of any DTaP-containing vaccines, receipt of the 4th dose of a Hib-containing vaccine, or receipt of the 3rd dose of PRP-OMP (PedvaxHIB® or Comvax® [Hep B-Hib]) prior to enrollment or during the conduction of the trial, except for Group 1 subjects, who may receive Hib vaccine at 12 months
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months). Topical steroids are not included in this exclusion criterion
* History of invasive meningococcal infection, confirmed either clinically, serologically, or microbiologically
* Personal history of Guillain-Barré Syndrome
* History of encephalopathy (e.g., coma, decreased level of consciousness, prolonged seizures) within 7 days of a previous dose of a pertussis containing vaccine that is not attributable to another identifiable cause
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to one of the vaccines used in the trial or to a vaccine containing any of the same substances
* Known thrombocytopenia, as reported by the parent/ legally acceptable representative, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* In an emergency setting or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/ infection (according to investigator judgment) or febrile illness (temperature ≥ 100.4°F [≥ 38.0°C]) on the day of vaccination. A prospective subject should not be included in the trial until the condition has resolved or the febrile event has subsided
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to any trial blood draw (topical antibiotics, drops, or ointments are not included in this criterion)
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed trial.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1394 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (55):
- United States (53):
  - Birmingham, Alabama
  - Pinson, Alabama
  - Tucson, Arizona
  - Fayetteville, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Chino, California
  - Downey, California
  - La Puente, California
  - Lakewood, California
  - Paramount, California
  - Norwich, Connecticut
  - Marietta, Georgia
  - Woodstock, Georgia
  - DeKalb, Illinois
  - Indianapolis, Indiana
  - Bossier City, Louisiana
  - Woburn, Massachusetts
  - Worcester, Massachusetts
  - Bridgeton, Missouri
  - Kansas City, Missouri
  - Elkhorn, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Clyde, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Fairfield, Ohio
  - Huber Heights, Ohio
  - Kettering, Ohio
  - Tulsa, Oklahoma
  - Erie, Pennsylvania
  - Harleysville, Pennsylvania
  - Hermitage, Pennsylvania
  - Scranton, Pennsylvania
  - Sellersville, Pennsylvania
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Hurst, Texas
  - San Antonio, Texas
  - Layton, Utah
  - Murray, Utah
  - Orem, Utah
  - Payson, Utah
  - Roy, Utah
  - Spanish Fork, Utah
  - Syracuse, Utah
  - Midlothian, Virginia
  - Spokane, Washington
- Puerto Rico (2):
  - Ponce, PR
  - San Juan, PR

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 24 July 2012 to 14 June 2013 in 62 clinical centers in the United States.
Pre-assignment Details: A total of 1394 participants were enrolled for the study, data on 1288 participants who met all the inclusion and none of the exclusion criteria and who completed the vaccination schedule are presented in this report.
Groups:
- Menactra Vaccine Group: All participants received Menactra vaccine at 9 months of age and a second dose of Menactra vaccine at age 15 to 18 months
- Menactra + Pentacel Vaccine Group: All participants received Menactra vaccine at 9 months of age and Menactra vaccine and Pentacel vaccine concomitantly at age 15 to 18 months.
- Pentacel Vaccine Group: Study participants received only Pentacel vaccine at 15 to 18 months of age
Period: Overall Study
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Started | 421 | 395 | 472
Completed | 413 | 388 | 461
Not Completed | 8 | 7 | 11
Not completed — Protocol Violation | 3 | 3 | 3
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 5

BASELINE CHARACTERISTICS:
Population: The demographic and baseline characteristics are in the safety analysis set (SafAS)
Groups:
- Menactra Vaccine Group: Study participants received Menactra vaccine at 9 months of age and a second dose of Menactra vaccine at age 15 to 18 months
- Menactra + Pentacel Vaccine Group: Study participants received Menactra vaccine at 9 months of age and Menactra vaccine and Pentacel vaccine concomitantly at age 15 to 18 months
- Total: Total of all reporting groups
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group | Total
Number analyzed (Participants) | 421 | 395 | 472 | 1288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 421 | 395 | 472 | 1288
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 284.5 (10.8) | 284.6 (10.6) | 483.9 (30.3) | 353.6 (96.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219 | 171 | 232 | 622
  Male | 202 | 224 | 240 | 666
Region of Enrollment [Number; unit: Participants]
  United States | 421 | 395 | 472 | 1288

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Study Participants Achieving Menactra Response for Meningococcal Serogroups A, C, Y, and W-135 Following the Second Menactra Vaccination
Description: Titers of antibodies to serogroups A, C, Y, and W-135 were measured by serum bactericidal assay using human complement (hSBA or SBA-HC).
  Menactra vaccine response defined as subjects with an hSBA titer <1:8 at baseline achieving an hSBA titer ≥1:8, and subjects with an hSBA titer ≥1:8 at baseline achieving a ≥ 4-fold increase in hSBA titer.
Time Frame: Day 30 post second Menactra vaccination
Population: Antibody titers to the meningococcal serogroups were assessed in the Per-protocol population of the participants in Menactra Vaccine Group and Menactra + Pentacel Vaccine Group.
Measure: Number; unit: Percentage of participants
Groups:
- Menactra Vaccine Group: Study participants that received Menactra vaccine at 9 months of age and a second dose of Menactra vaccine at age 15 to 18 months.
- Menactra + Pentacel Vaccine Group: Study participants that received Menactra vaccine at 9 months of age and Menactra vaccine and Pentacel vaccine concomitantly at age 15 to 18 months.
- Pentacel Vaccine Group: Study participants that received only Pentacel vaccine at 15 to 18 months of age
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 352 | 333 | 0
Percentage of participants
  Serogroup A (N=346, 329, 0) | 96.24 | 96.35 |
  Serogroup C (N=352, 333, 0) | 98.86 | 97.60 |
  Serogroup Y (N=351, 333, 0) | 98.86 | 96.40 |
  Serogroup W-135 (N=351, 330, 0) | 98.86 | 97.58 |
Statistical Analysis 1: Comparison: Menactra Vaccine Group vs Menactra + Pentacel Vaccine Group; Meningococcal serogroup A: The null hypothesis (H0: pm - ppm > δ) was tested against the alternative hypothesis (H1: pm - ppm ≤ δ), where pm and ppm were the proportions of subjects in Group 1 and in Group 2, respectively, who achieved a Menactra vaccine response for meningococcal serogroups A, C, Y and W-135, with δ = 0.10; Test type: Non-Inferiority or Equivalence — If the upper limit of the two-sided 95% confidence interval (CI) of the difference between the two proportions was < δ for serogroup A and assuming the difference between the two proportions was normally distributed, the inferiority assumption was to be rejected; Difference between 2 percentages = -0.110, 95% CI 2-sided [-3.11 to 2.93]
Statistical Analysis 2: Comparison: Menactra Vaccine Group vs Menactra + Pentacel Vaccine Group; Meningococcal serogroup C: The null hypothesis (H0: pm - ppm > δ) was tested against the alternative hypothesis (H1: pm - ppm ≤ δ), where pm and ppm were the proportions of subjects in Group 1 and in Group 2, respectively, who achieved a Menactra vaccine response for meningococcal serogroups A, C, Y and W-135, with δ = 0.10; Test type: Non-Inferiority or Equivalence — If the upper limit of the two-sided 95% CI of the difference between the two proportions was < δ for serogroup C and assuming the difference between the two proportions was normally distributed, the inferiority assumption was to be rejected; Difference between 2 percentages = 1.27, 95% CI 2-sided [-0.84 to 3.64]
Statistical Analysis 3: Comparison: Menactra Vaccine Group vs Menactra + Pentacel Vaccine Group; Meningococcal serogroup Y: The null hypothesis (H0: pm - ppm > δ) was tested against the alternative hypothesis (H1: pm - ppm ≤ δ), where pm and ppm were the proportions of subjects in Group 1 and in Group 2, respectively, who achieved a Menactra vaccine response for meningococcal serogroups A, C, Y and W-135, with δ = 0.10; Test type: Non-Inferiority or Equivalence — If the upper limit of the two-sided 95% CI of the difference between the two proportions was < δ for serogroup Y and assuming the difference between the two proportions was normally distributed, the inferiority assumption was to be rejected; Difference between 2 percentages = 2.46, 95% CI 2-sided [0.14 to 5.14]
Statistical Analysis 4: Comparison: Menactra Vaccine Group vs Menactra + Pentacel Vaccine Group; Meningococcal serogroup W-135: The null hypothesis (H0: pm - ppm > δ) was tested against the alternative hypothesis (H1: pm - ppm ≤ δ), where pm and ppm were the proportions of subjects in Group 1 and in Group 2, respectively, who achieved a Menactra vaccine response for meningococcal serogroups A, C, Y and W-135, with δ = 0.10; Test type: Non-Inferiority or Equivalence — If the upper limit of the two-sided 95% CI of the difference between the two proportions was < δ for serogroup W-135 and assuming the difference between the two proportions was normally distributed, the inferiority assumption was to be rejected; Difference between 2 percentages = 1.28, 95% CI 2-sided [-0.84 to 3.67]

2. Other Pre Specified Outcome: Geometric Mean Titers of Individual Meningococcal Antibodies in Serum Bactericidal Assay With Human Complement (SBA-HC) Analysis Following Vaccination With Menactra Vaccine
Description: Geometric mean titers (GMTs) of antibodies to serogroups A, C, Y, and W-135 were measured by serum bactericidal assay with human complement (SBA HC) before any vaccination and post-vaccination 2
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination 2
Population: Geometric mean titers of individual antibodies were assessed in the Per-protocol population in the Menactra Vaccine Group and Menactra + Pentacel Vaccine Group participants.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 356 | 336 | 0
Titers
  Serogroup A (Pre-vaccination; N=352, 332, 0) | 3.4 [3.16 to 3.74] | 4.3 [4.01 to 4.54] |
  Serogroup A (Post-vaccination; N=350, 332, 0) | 104.8 [91.6 to 120] | 104.5 [90.9 to 120] |
  Serogroup C (Pre-vaccination; N=352, 332, 0) | 2.2 [2.10 to 2.23] | 2.1 [2.03 to 2.16] |
  Serogroup C (Post-vaccination; N=350, 332, 0) | 157.9 [139 to 179] | 129.1 [113 to 148] |
  Serogroup Y (Pre-vaccination; N=352, 332, 0) | 2.1 [2.02 to 2.12] | 2.1 [2.03 to 2.17] |
  Serogroup Y (Post-vaccination; N=350, 332, 0) | 77.8 [69.3 to 87.4] | 62.2 [54.7 to 70.7] |
  Serogroup W-135 (Pre-vaccination; N=352, 332, 0) | 2.1 [2.05 to 2.13] | 2.1 [2.01 to 2.13] |
  Serogroup W-135 (Post-vaccination; N=350, 332, 0) | 90.3 [78.9 to 103] | 81.1 [70.9 to 92.8] |

3. Other Pre Specified Outcome: Geometric Mean Titers of Individual Antibodies to Filamentous Hemagglutinin, Pertactin, Diphtheria, Tetanus and Polio Antigens Following Vaccination With Either Pentacel Only or Menactra Concomitantly With Pentacel Vaccine
Description: Filamentous hemagglutinin (FHA), Fimbriae types 2 and 3 (FIM), Pertactin (PRN) and anti-Tetanus antibodies were measured by enzyme-linked immunosorbent assay (ELISA); anti-Diphtheria antibodies were measured by a toxin neutralization test.
Time Frame: Day 0 (pre-vaccination) and Day 30 post-vaccination 2
Population: Geometric mean titers of individual vaccine antibodies were assessed in the Per-protocol population of the Menactra + Pentacel Vaccine Group and the Pentacel Vaccine Group participants.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 0 | 336 | 418
Titers
  Anti-FIM (pre-vaccination; N=0, 335, 418) |  | 17.6 [15.5 to 19.8] | 23.2 [20.8 to 25.9]
  Anti-FIM (post-vaccination; N=0, 332, 417) |  | 220.8 [191 to 255] | 265.5 [233 to 302]
  Anti-PRN (pre-vaccination; N=0, 334, 418) |  | 10.3 [9.18 to 11.6] | 11.1 [9.95 to 12.3]
  Anti-PRN (post-vaccination; N=0, 331, 417) |  | 120.9 [107 to 137] | 133.9 [120 to 150]
  Anti-Diphtheria (pre-vaccination; N=0, 328, 418) |  | 0.3 [0.235 to 0.306] | 0.2 [0.179 to 0.225]
  Anti-Diphtheria (post-vaccination; N=0, 324, 416) |  | 3.3 [3.00 to 3.68] | 4.2 [3.85 to 4.54]
  Anti-Tetanus (pre-vaccination; N=0, 329, 414) |  | 0.2 [0.2 to 0.268] | 0.2 [0.2 to 0.267]
  Anti-Tetanus (post-vaccination; N=0, 326, 415) |  | 3.7 [3.38 to 3.99] | 3.9 [3.56 to 4.18]
  Anti-Polio 1 (pre-vaccination; N=0, 326, 415) |  | 83.1 [70.4 to 98.0] | 76.9 [64.7 to 91.2]
  Anti-Polio 1 (post-vaccination; N=0, 323, 414) |  | 2140 [1819 to 2518] | 1887 [1653 to 2153]
  Anti-Polio 2 (pre-vaccination; N=0, 328, 417) |  | 157.0 [136 to 181] | 182.8 [157 to 212]
  Anti-Polio 2 (post-vaccination; N=0, 324, 414) |  | 3172 [2800 to 3593] | 3071 [2754 to 3425]
  Anti-Polio 3 (pre-vaccination; N=0, 327, 417) |  | 107.1 [90.7 to 127] | 130.2 [110 to 155]
  Anti-Polio 3 (post-vaccination; N=0, 323, 415) |  | 4629 [3980 to 5384] | 3765 [3305 to 4288]

4. Other Pre Specified Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reactions Following Vaccination With Menactra Only, or Pentacel Only or Menactra Concomitantly With Pentacel Vaccine
Description: Solicited injection-site reactions: Tenderness, Erythema, and Swelling. Solicited Systemic Reactions: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite, and Irritability. Grade 3 solicited reactions defined as: Tenderness - cries when injected limb is moved, or the movement of the injected limb is reduced; Erythema and Swelling - ≥ 50 mm; Fever > 39.5°C or > 103.1 °F; Vomiting - ≥ 6 episodes per 24 hours or requiring parenteral hydration; Abnormal crying > 3 hours; Drowsiness - Sleeping most of the time or difficult to wake up; Loss of appetite - Refuses ≥ 3 feeds / meals or refuses most feeds / meals; and Irritability - Inconsolable.
Time Frame: Day 0 to Day 7 after any vaccination
Population: Solicited reactions were assessed in all subjects who received at least one dose of study vaccine, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 421 | 395 | 472
Percentage of participants
  Any injection-site Tenderness (N = 420, 393, 463) | 52.1 | 61.6 | 51.4
  Grade 3 inj.-siteTenderness (N = 420, 393, 463) | 1.0 | 4.3 | 1.9
  Any injection-site Erythema (N = 420, 393, 463) | 25.2 | 38.7 | 31.1
  Grade 3 inj.-site Erythema (N = 420, 393, 463) | 0.2 | 0.8 | 1.1
  Any injection-site Swelling (N = 420, 393, 463) | 15.0 | 23.2 | 21.4
  Grade 3 inj.-site Swelling (N = 420, 393, 463) | 0.0 | 0.3 | 0.6
  Any Fever (N = 421, 394, 463) | 16.9 | 21.6 | 12.3
  Grade 3 Fever (N = 421, 394, 463) | 1.4 | 2.8 | 0.9
  Any Vomiting (N = 420, 393, 463) | 22.6 | 17.3 | 9.9
  Grade 3 Vomiting (N = 420, 393, 463) | 0.5 | 0.3 | 0.6
  Any Crying abnormal (N = 420, 393, 463) | 52.9 | 52.2 | 39.1
  Grade 3 Crying abnormal (N = 420, 393, 463) | 4.0 | 5.1 | 2.2
  Any Drowsiness (N = 420, 393, 463) | 49.8 | 52.4 | 30.0
  Grade 3 Drowsiness (N = 421, 394, 463) | 3.1 | 2.0 | 1.7
  Appetite lost (N = 420, 393, 463) | 43.3 | 47.8 | 35.2
  Grade 3 Appetite lost (N = 420, 393, 463) | 2.1 | 3.3 | 1.3
  Any Irritability (N = 420, 393, 463) | 70.5 | 72.3 | 58.5
  Grade 3 Irritability (N = 420, 393, 463) | 6.4 | 6.9 | 2.4

5. Other Pre Specified Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reactions Following Vaccination at 9 Months of Age With Menactra Vaccine.
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited Systemic Reactions: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite, and Irritability. Grade 3 solicited reactions defined as: Tenderness - cries when injected limb is moved, or the movement of the injected limb is reduced; Erythema and Swelling - ≥ 50 mm; Fever > 39.5°C or > 103.1 °F; Vomiting - ≥ 6 episodes per 24 hours or requiring parenteral hydration; Abnormal crying > 3 hours; Drowsiness - Sleeping most of the time or difficult to wake up; Loss of appetite - Refuses ≥ 3 feeds / meals or refuses most feeds/meals; and Irritability - Inconsolable.
Time Frame: Day 0 to Day 7 after 9-month vaccination
Population: Solicited reactions were assessed in subjects who received at least one dose of study vaccine at 9 month of age, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 421 | 395 | 0
Percentage of participants
  Any injection-site Tenderness (N = 419, 387, 0) | 32.2 | 34.1 |
  Grade 3 injection-site Tenderness (N=419, 387, 0) | 0.2 | 0.8 |
  Any injection-site Erythema (N = 419, 387, 0) | 16.9 | 24.3 |
  Grade 3 injection-site Erythema (N = 419, 387, 0) | 0.0 | 0.0 |
  Any injection-site Swelling (N = 419, 385, 0) | 10.0 | 9.4 |
  Grade 3 injection-site Swelling (N = 419, 385, 0) | 0.0 | 0.0 |
  Any Fever (N = 421, 389, 0) | 10.5 | 10.3 |
  Grade 3 Fever (N = 421, 389, 0) | 0.7 | 1.5 |
  Any Vomiting (N = 419, 387, 0) | 15.5 | 12.9 |
  Grade 3 Vomiting (N = 419, 387, 0) | 0.5 | 0.0 |
  Any Crying abnormal (N = 419, 387, 0) | 38.9 | 37.5 |
  Grade 3 Crying abnormal (N = 419, 387, 0) | 3.3 | 2.8 |
  Any Drowsiness (N = 419, 387, 0) | 37.2 | 37.0 |
  Grade 3 Drowsiness (N = 419, 387, 0) | 2.1 | 0.8 |
  Appetite lost (N = 419, 387, 0) | 25.3 | 28.7 |
  Grade 3 Appetite lost (N = 419, 387, 0) | 1.4 | 1.8 |
  Any Irritability (N = 419, 387, 0) | 56.1 | 54.8 |
  Grade 3 Irritability (N = 419, 387, 0) | 4.8 | 3.1 |

6. Primary Outcome: Geometric Mean Concentrations of Pertussis Vaccine Antibodies Following Vaccination With Either Pentacel Only or Menactra Concomitantly With Pentacel Vaccine
Description: Pertussis antibodies, anti-Pertussis toxoid (PT), Filamentous hemagglutinin (FHA), Pertactin (PRN) antibodies were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 30 post-vaccination 2
Population: Geometric Mean Concentrations (GMC) of Pertussis vaccine antibodies were assessed in the Per-protocol population of participants in Menactra + Pentacel Vaccine Group and Pentacel Vaccine Group.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 0 | 332 | 417
Titers
  Anti-Pertussis Toxoid (PT; N=0, 332, 417) |  | 73.5 [67.9 to 79.6] | 69.7 [64.9 to 75.0]
  Anti-Filamentous hemagglutinin FHA; N=0, 331, 417) |  | 113.7 [105 to 123] | 110.1 [102 to 119]
  Anti-Pertactin (PRN; N=0, 331, 417) |  | 120.9 [107 to 137] | 133.9 [120 to 150]
Statistical Analysis 1: Comparison: Menactra + Pentacel Vaccine Group vs Pentacel Vaccine Group; Pertussis toxoid (PT): The null hypothesis (H0: GMCp / GMCpm > 1.5) was tested against the alternative hypothesis (H1: GMCp / GMCpm ≤ 1.5), where GMCp and GMCpm were the GMCs of antibodies against the pertussis antigen (PT) in Group 3 and in Group 2, respectively; Test type: Non-Inferiority or Equivalence — Assuming that the antibodies concentration was log normally distributed, if the upper limit of the two-sided 95% CI of the ratio of the two GMCs is ≤ 1.5 for each antigen, the inferiority assumption was to be rejected; Mean Difference (Final Values) = 0.949, 95% CI 2-sided [0.852 to 1.06]
Statistical Analysis 2: Comparison: Menactra + Pentacel Vaccine Group vs Pentacel Vaccine Group; Filamentous hemagglutinin (FHA): The null hypothesis (H0: GMCp / GMCpm > 1.5) was tested against the alternative hypothesis (H1: GMCp / GMCpm ≤ 1.5), where GMCp and GMCpm were the GMCs of antibodies against the pertussis antigen (FHA) in Group 3 and in Group 2, respectively; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.968, 95% CI 2-sided [0.866 to 1.08]
Statistical Analysis 3: Comparison: Menactra + Pentacel Vaccine Group vs Pentacel Vaccine Group; Pertactin (PRN): The null hypothesis (H0: GMCp / GMCpm > 1.5) was tested against the alternative hypothesis (H1: GMCp / GMCpm ≤ 1.5), where GMCp and GMCpm were the GMCs of antibodies against the pertussis antigen (PRN) in Group 3 and in Group 2, respectively; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [0.937 to 1.31]

7. Primary Outcome: Percentage of Participants With Pertussis Vaccine Responses Following Vaccination With Either Pentacel Only or Menactra Concomitantly With Pentacel Vaccine
Description: Pertussis antibodies, anti-Pertussis toxoid (PT), Filamentous hemagglutinin (FHA), and Pertactin (PRN) antibodies were measured by enzyme-linked immunosorbent assay (ELISA). Pertussis response was defined as: ≥4 × baseline concentration, if the anti-pertussis antibody concentration at baseline is <4 × lower limit of quantification (LLOQ), Or ≥2 × baseline concentration, if the anti-pertussis antibody concentration at baseline is ≥4 × LLOQ
Time Frame: Day 30 post-vaccination 2
Population: Antibody responses to Pertussis vaccine antigens were assessed in the Per-protocol population of the Menactra + Pentacel Vaccine Group and Pentacel Vaccine Group participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 0 | 330 | 417
Percentage of Participants
  Anti-Pertussis Toxoid (PT; N=0, 330, 417) |  | 90.91 | 89.69
  Anti-Filamentous hemagglutinin (FHA; N=0,329, 417) |  | 93.62 | 94.48
  Anti-Pertactin (PRN; N=0, 329, 417) |  | 93.62 | 93.53
Statistical Analysis 1: Comparison: Menactra + Pentacel Vaccine Group vs Pentacel Vaccine Group; Pertussis toxoid (PT) antigen: The null hypothesis (H0: pp - ppm > δ) was tested against the alternative hypothesis (H1: pp - ppm ≤ δ), where pp and ppm were the proportions of subjects in Group 3 and Group 2, respectively, who achieved a pertussis vaccine response in antibodies against the pertussis antigen (PT), with δ = 0.10; Test type: Non-Inferiority or Equivalence — If the upper limit of the two-sided 95% CI of the difference between the two proportions was < δ for each antibody and assuming the difference between the two proportions was normally distributed, the inferiority assumption was to be rejected; Difference between 2 percentages = -1.22, 95% CI 2-sided [-5.44 to 3.19]
Statistical Analysis 2: Comparison: Menactra + Pentacel Vaccine Group vs Pentacel Vaccine Group; Filamentous hemagglutinin (FHA) antigen: The null hypothesis (H0: pp - ppm > δ) was tested against the alternative hypothesis (H1: pp - ppm ≤ δ), where pp and ppm were the proportions of subjects in Group 3 and Group 2, respectively, who achieved a pertussis vaccine response in antibodies against the pertussis antigen (FHA), with δ = 0.10; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; Difference between 2 percentages = 0.867, 95% CI 2-sided [-2.54 to 4.53]
Statistical Analysis 3: Comparison: Menactra + Pentacel Vaccine Group vs Pentacel Vaccine Group; Pertactin (PRN) antigen: The null hypothesis (H0: pp - ppm > δ) was tested against the alternative hypothesis (H1: pp - ppm ≤ δ), where pp and ppm were the proportions of subjects in Group 3 and Group 2, respectively, who achieved a pertussis vaccine response in antibodies against the pertussis antigen (PRN), with δ = 0.10; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 7, analysis 1]; Difference between 2 percentages = -0.092, 95% CI 2-sided [-3.62 to 3.66]

8. Other Pre Specified Outcome: Percentage of Participants Reporting Solicited Injection-site or Systemic Reactions Following Vaccination With Menactra Only, or Pentacel Only, or Menactra Concomitantly With Pentacel Vaccine
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite, and Irritability. Grade 3 reactions defined as: Tenderness - cries when injected limb is moved, or the movement of the injected limb is reduced; Erythema and Swelling - ≥ 50 mm; Fever > 39.5°C or > 103.1 °F; Vomiting - ≥ 6 episodes per 24 hours or requiring parenteral hydration; Abnormal crying > 3 hours; Drowsiness - Sleeping most of the time or difficult to wake up; Loss of appetite - Refuses ≥ 3 feeds/meals or refuses most feeds/meals; and Irritability - Inconsolable.
Time Frame: Day 0 to Day 7 after the 15 to 18 month vaccination
Population: Solicited reactions were assessed in all subjects who received at least one dose of 15 to 18 month study vaccine, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Percentage of participants
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 421 | 395 | 472
Percentage of participants
  Any injection-site Tenderness (N = 411, 382, 463) | 37.0 | 54.7 | 51.4
  Grade 3 inj.-site Tenderness (N = 411, 382, 463) | 0.7 | 3.7 | 1.9
  Any injection-site Erythema (N = 411, 382, 463) | 17.8 | 30.1 | 31.1
  Grade 3 injection-site Erythema (N=411, 382, 463) | 0.2 | 0.8 | 1.1
  Any injection-site Swelling (N = 411, 382, 463) | 9.2 | 19.6 | 21.4
  Grade 3 injection-site Swelling (N=411, 382, 463) | 0.0 | 0.3 | 0.6
  Any Fever (N = 412, 385, 463) | 8.5 | 14.3 | 12.3
  Grade 3 Fever (N = 412, 385, 463) | 0.7 | 1.3 | 0.9
  Any Vomiting (N = 411, 382, 463) | 10.0 | 7.9 | 9.9
  Grade 3 Vomiting (N = 411, 382, 463) | 0.0 | 0.3 | 0.6
  Any Crying abnormal (N = 411, 382, 463) | 33.8 | 37.2 | 39.1
  Grade 3 Crying abnormal (N = 411, 382, 463) | 1.0 | 2.6 | 2.2
  Any Drowsiness (N = 411, 382, 463) | 30.9 | 40.6 | 30.0
  Grade 3 Drowsiness (N = 411, 382, 463) | 1.0 | 1.3 | 1.7
  Appetite lost (N = 411, 382, 463) | 29.7 | 34.0 | 35.2
  Grade 3 Appetite lost (N = 411, 382, 463) | 0.7 | 1.6 | 1.3
  Any Irritability (N = 411, 382, 463) | 50.6 | 57.9 | 58.5
  Grade 3 Irritability (N = 411, 382, 463) | 2.7 | 3.9 | 2.4

9. Primary Outcome: Percentage of Participants With Antibody Responses to Diphtheria, Tetanus and Polyribosylribitol Phosphate Antigens Following Vaccination With Either Pentacel Only or Menactra Concomitantly With Pentacel Vaccine
Description: Anti-Tetanus antibodies were measured by enzyme-linked immunosorbent assay (ELISA), anti-polyribosylribitol phosphate (PRP) antibodies were measured using a Farr-type radioimmunoassay, and anti-diphtheria antibodies were measured by a toxin neutralization test.
  The vaccine responses were defined as: Anti-PRP antibody concentrations ≥1.0 μg/mL; Anti-tetanus antibody concentrations ≥1.0 IU/mL and Anti-diphtheria antibody concentrations ≥1.0 IU/mL, respectively, 30 days after vaccination with Pentacel® in participants in Groups 2 and 3.
Time Frame: Day 30 post-vaccination 2
Population: Antibody responses to Diphtheria, Tetanus, and Polyribosylribitol phosphate antigens were assessed in the Per-protocol population of the Menactra + Pentacel Vaccine Group and Pentacel Vaccine Group participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Number analyzed (Participants) | 0 | 336 | 418
Percentage of Participants
  Anti-Diphtheria (N=0, 324, 416) |  | 99.69 | 100.00
  Anti-Tetanus (N=0, 326, 415) |  | 100.00 | 100.00
  Anti-Polyribosylribitol phosphate (N=0, 324, 416) |  | 97.53 | 97.12

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from vaccination on Day 0 through Day 30 post-second (final) vaccination.
Arm/Group | Menactra Vaccine Group | Menactra + Pentacel Vaccine Group | Pentacel Vaccine Group
Serious Adverse Events (participants affected / at risk) | 13/421 | 11/395 | 1/472
Other Adverse Events (participants affected / at risk) | 296/421 | 318/395 | 380/472
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra Vaccine Group (N=421) | Menactra + Pentacel Vaccine Group (N=395) | Pentacel Vaccine Group (N=472)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Penile abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Menactra Vaccine Group (N=421) | Menactra + Pentacel Vaccine Group (N=395) | Pentacel Vaccine Group (N=472)
Injection Site Tenderness (General disorders) | 219/420 (219) | 242/393 (242) | 238/463 (238)
Injection Site Erythema (General disorders) | 106/420 (106) | 152/393 (152) | 144/463 (144)
Vomiting (Gastrointestinal disorders) | 95/420 (95) | 68/393 (68) | 46 (46)
Fever (General disorders) | 71 (71) | 85/394 (85) | 57/463 (57)
Crying abnormal (Psychiatric disorders) | 222/420 (222) | 205/393 (205) | 181/463 (181)
Drowsiness (Nervous system disorders) | 209/420 (209) | 206/393 (206) | 139/463 (139)
Appetite lost (Metabolism and nutrition disorders) | 182/420 (182) | 188/393 (188) | 163/463 (163)
Diarrhoea (Gastrointestinal disorders) | 30 (35) | 21 (22) | 26 (29)
Teething (Gastrointestinal disorders) | 31 (39) | 24 (33) | 42 (47)
Pyrexia (General disorders) | 42 (47) | 36 (40) | 25 (27)
Otitis media (Infections and infestations) | 58 (69) | 50 (57) | 28 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 60 (66) | 44 (48) | 31 (31)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 43 (48) | 47 (54) | 22 (22)
Upper respiratory tract infection (Infections and infestations) | 60 (64) | 52 (58) | 50 (51)
Injection-site Swelling (General disorders) | 63/420 (63) | 91/393 (91) | 99/463 (99)
Irritability (Psychiatric disorders) | 296/420 (296) | 284/393 (284) | 271/463 (271)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications